CLINICAL TRIAL: NCT06521008
Title: Effect of Diaphragmatic Training on Urgency Urinary Incontinence in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sandy Samir Hassan Darweesh, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sandy PHD
Record Dates: First submitted 2024-06-30; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Urge Incontinence; Urinary Incontinence; Postmenopausal Disorder
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: single blinded randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Selctive drugs (Experimental): consists of 20 women. They will receive selective anti Muscarinic drugs (5-10 mg) once per day for 12 weeks and instructions including bladder retraining.
  Interventions: Drug: anti muscarinic drugs; Other: Instructions including bladder training
- Pelvic floor and abdominal strengthening (Experimental): consists of 20 women. They will receive the same treatment in group (A), pelvic floor muscle training (PFMT) and abdominal strengthening 3 sessions/week for 12 weeks.
  Interventions: Drug: anti muscarinic drugs; Other: Instructions including bladder training; Other: pelvic floor muscle training (PFMT); Other: abdominal exercise
- diaphragmatic training (Experimental): consists of 20 women. They will receive the same treatment in group (B), in addition to diaphragmatic training 3 sessions/week for 12 weeks.
  Interventions: Drug: anti muscarinic drugs; Other: Instructions including bladder training; Other: Diaphragmatic Training

INTERVENTIONS:
Drug: anti muscarinic drugs — a selective anti muscarinic drugs (5-10mg) once per day for 12 weeks.
Other: Instructions including bladder training — The program teaches women skills and strategies to prevent incontinence, including bladder irritants like caffeine and discussing bowel habits to prevent constipation. It also teaches them how to respond adaptively to urgency, such as pause, sit down, relax, and contract pelvic muscles to diminish urgency and prevent urine loss. Once urgency subsides, they can proceed to the toilet at a normal pace. The program emphasizes the importance of educating patients about bladder irritants and bowel habits.
Other: pelvic floor muscle training (PFMT) — The training program teaches bladder control through contracting the striated skeletal pelvic floor muscles (PFM). The women are instructed to empty their bladder, lie in a lithotomy position, and tighten their pelvic floor muscles. The duration of contraction and repetitions is gradually increased, totaling 20-30 minutes. The program is 3 sessions per week under supervision for 12 weeks, and each woman is instructed to perform exercises at home until they can do 300 contractions per day.
  Arms: Pelvic floor and abdominal strengthening
Other: abdominal exercise — Women will engage in transverse abdominis exercises, focusing on drawing the lower abdominal wall towards the spine and pressing the lumbar region downward, repeated for 15 minutes per session, three times per week.
  Arms: Pelvic floor and abdominal strengthening
Other: Diaphragmatic Training — The therapist will instruct each woman to lie on her back with knees bent, place one hand on her upper chest and the other on her belly. They will breathe in slowly, tighten abdominal muscles, and exhale through pursed lips. Expiration should be relaxed and lightly controlled, and not forceful. Expiration should not be prolonged, and the woman should not initiate inspiration with accessory muscles or upper chest. The session will be repeated 3-4 times, lasting 5-10 minutes, and repeated three times per week for 12 weeks.
  Arms: diaphragmatic training

SUMMARY:
The purpose of this study was to determine the effect of diaphragmatic training on urgency urinary incontinence in postmenopausal women.

DETAILED DESCRIPTION:
Urgency urinary incontinence affects 9-13% of women, increasing with age and impacting daily activities, quality of life, depression, and social isolation. It is a significant source of dependency among the elderly and a factor in nursing home admissions. Untreated incontinence can lead to falls, infections, and loss of independence. Conservative management is the first-line therapy, but pelvic floor muscle training is a potential treatment method. This study aims to evaluate the effectiveness of diaphragmatic training on urinary incontinence in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women suffer from UUI.
* They will be multipara more than 1.
* Their age will range from 55-65 years old.
* Their body mass index (BMI) will range from 25-29.9 kg/m2..
* They will experience menopause at least for 3 years.

Exclusion Criteria:

* Urinary tract infection
* Previous surgery for urinary incontinence
* Upper motor neuron diseases
* History of genito-urinary cancer
* Previous pelvic irradiation
* Pure stress urinary incontinence
* Genital prolapse
* Diabetes mellitus
* Pace maker

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women suffer from Urgency urinary incontinence
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
assessing the change in Urodynamics (first desire to void) | up to 12 weeks
  The study used a double-lumen cytometry catheter to diagnose involuntary detrusor contractions in women. The catheter measured the change in urodynamics in form of volume at first desire to void, for each woman in all groups. The urodynamic method is a reliable and mandatory method for diagnosing and treating UUI symptoms, as relying solely on urinary symptoms may lead to under-diagnosis of detrusor overactivity.
assessing the change in Urodynamics (first sensation of bladder filling) | up to 12 weeks
  The study used a double-lumen cytometry catheter to diagnose involuntary detrusor contractions in women. The catheter measured the change in urodynamics in form of first sensation of bladder filling, for each woman in all groups.
assessing the change in Urodynamics (maximum bladder capacity) | up to 12 weeks
  The study used a double-lumen cytometry catheter to diagnose involuntary detrusor contractions in women. The catheter measured the change in urodynamics in form of maximum bladder capacity, for each woman in all groups.

SECONDARY OUTCOMES:
assessing the change in weight and height | up to 12 weeks
  The study utilized a weight-height scale to measure weight and height for women in all groups (A, B & C) and to calculate BMI before and after treatment.
assessing the change in bladder ascending movement | up to 12 weeks
  Transvaginal ultrasound assessment of bladder and urethra was conducted in the midsagittal plane, determining posterior urethro vesical angle.
assessing the change in Urinary function | up to 12 weeks
  The study uses a self-administered questionnaire to assess urinary function in women in different groups (A, B, and C) at the start and end of the study course. The questionnaire consists of 21 items, each with its own Likert rating scale structure. Each woman is instructed and given appropriate time to answer.
assessing the change in body mass index | up to 12 weeks
  The study utilized a weight-height scale to measure to calculate BMI before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- OM El Masreen General Hospital, Giza, Egypt